CLINICAL TRIAL: NCT07030114
Title: Impact of Mechanical Ventilation on Hematological Parameters in Pediatric Patients With Sepsis
Brief Title: The Study Seeks to Determine Potential Correlations Between Ventilation and Hematological Alterations, Contributing to a Better Understanding of Its Physiological Effects and Optimizing Patient Management in Critical Care Settings.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Magdy Abdelazeem Ahmed, Principal Investigator, Assiut University
Other Study IDs: hematology and MV in sepsis
Record Dates: First submitted 2025-05-05; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Sepsis-induced Multiple Organ Dysfunction Syndrome
Keywords: hematological changes; lab investigation; pediatric patients; sepsis; mechanical ventilation
MeSH Terms: conditions — Sepsis | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: complete blood tests — Complete Blood Count (CBC): Using automated hematology analyzers to measure various blood cell parameters.
  * C-Reactive Protein (CRP): Quantitative analysis using immunoturbidimetric assay.
  * Erythrocyte Sedimentation Rate (ESR): Measured using the Westergren method.
  * Coagulation profile:
  * Prothrombin Time (PT): Using thromboplastin reagents and automated coagulation analyzers.
  * Activated Partial Thromboplastin Time (aPTT): Using phospholipid-based reagents and automated analyzers.
  * International Normalized Ratio (INR): Calculated from PT results.
  * Bleeding Time: Ivy method or template bleeding time.
  * Liver function tests: Including ALT, AST, ALP, bilirubin using spectrophotometric methods.
  * Kidney function tests: Creatinine and BUN using enzymatic methods.
Device: mechanical ventilation (MV) — Mechanical Ventilation Parameters
  * - Ventilation Mode: Ventilator settings will record modes such as volume-controlled ventilation or synchronized intermittent mandatory ventilation (SIMV), which deliver breaths based on patient needs.
  * Tidal Volume: Measured in milliliters per kilogram of predicted body weight. Tidal volume settings aim to optimize oxygenation while minimizing lung injury risks by adhering to evidence-based limits (<6 mL/kg).
  * Positive End-Expiratory Pressure (PEEP): PEEP levels will be recorded in cmH₂O to prevent alveolar collapse and improve oxygenation. Adjustments will balance oxygenation benefits with potential risks like reduced venous return or lung overdistension.
  * Fraction of Inspired Oxygen (FiO₂): FiO₂ values will be documented as decimals, starting at 1.0 (100% oxygen) and adjusted downward based on patient oxygenation needs.

SUMMARY:
The study seeks to determine potential correlations between ventilation and hematological alterations, contributing to a better understanding of its physiological effects and optimizing patient management in critical care settings.

DETAILED DESCRIPTION:
* Sepsis is a clinical disorder caused by a dysregulated host response to severe infection. Pediatric sepsis remains a major public health issue and a significant cause of morbidity and mortality despite the development of standardized treatment guidelines, universal immunization programs, and advanced intensive-care organ support techniques. Severe sepsis is responsible for > 8% of all pediatric intensive care unit (PICU) admissions and causes > 4.5 million childhood deaths worldwide per year.
* However, the clinical manifestations of these infections vary from minimal symptoms to multiple organ failure and death. The currently accepted definitions of sepsis, severe sepsis, and septic shock were developed and refined using different criteria to help identify, treat, and study patients with infections who are at higher risk of significant morbidity and mortality as it is responsible of 25% of deaths in children worldwide.
* The onset, progression and outcome of sepsis are frequently associated with coagulation abnormalities, and the excessive crosstalk between inflammation and coagulation plays a vital role in these pathogenesis, which includes dysfunction of clotting cascade process, anticoagulant and fibrinolytic systems, together with related endothelial damage. Sepsis-related coagulopathy can range in severity from mildly decreased platelet counts and prolonged clotting time, which are indicative of subclinical issues, to more severe coagulopathies such as disseminated intravascular coagulation (DIC). Classic coagulation laboratory tests, such as activated partial thromboplastin time (APTT), prothrombin time (PT), and platelet count, mainly indicate signs of consumption and impaired synthesis instead of ongoing coagulopathy and change slowly in the disease course .
* Mechanical ventilation (MV) is a common practice in pediatric intensive care units (PICUs). Its utilization rate, as reported in multicenter and prospective studies in heterogeneous cohorts, varies from 20% to 50% of the patients admitted to these units. Mechanical ventilation is a crucial intervention in pediatric intensive care units (PICUs), particularly for children with sepsis. Sepsis, a life-threatening condition resulting from an uncontrolled immune response to infection, often necessitates invasive mechanical ventilation (IMV) to manage respiratory failure and maintain adequate blood gas levels. The duration of mechanical ventilation can significantly impact patient outcomes, with prolonged use associated with increased risks of complications such as ventilator-associated pneumonia (VAP) and longer hospital stays.
* Accurate and early diagnosis is important to initiate effective treatment and improve the prognosis of sepsis. Therefore, a large number of biomarkers have been developed to diagnose sepsis. Unfortunately, none of these biomarkers exhibit a high degree of sensitivity and specificity. The most common of these markers is C-reactive protein (CRP), which is a major acute-phase reactant in infection and inflammation.
* CBC is an inexpensive, simple, routine, and repeatable test used to indicate the presence of infection. Leucocyte numbers and neutrophil ratios were the most commonly used indices for detecting infections. Recently, other CBC parameters, such as NLR and PLR, have been used in children and adult patients to identify inflammatory processes. These parameters are routinely measured in all patients admitted to the PICU.
* The collaboration between mechanical ventilation and hematological parameters in pediatric sepsis patients is an area that warrants thorough investigation. Hematological abnormalities, including anemia, thrombocytopenia, and coagulopathies, are prevalent in sepsis and can adversely affect patient outcomes. Understanding how MV influences these parameters is essential for optimizing treatment protocols and improving prognoses. Despite the high incidence of MV in Egyptian PICUs, there is a gap in research focusing on its impact on hematological profiles in this demographic. Addressing this gap could lead to enhanced clinical practices and better patient outcomes in pediatric sepsis care.

ELIGIBILITY:
Inclusion Criteria:

* 1- Pediatric patients aged 1 month to 18 years 2- Diagnosis of sepsis based on (Specify Criteria, e.g., Sepsis-3 criteria) 3- Requirement for invasive mechanical ventilation for at least 24 hours. 4- Patients admitted to the PICU during the study period. 5- Availability of complete hematological data before and during mechanical ventilation

Exclusion Criteria:

* 1- Patients with pre-existing hematological disorders (e.g., leukemia, aplastic anemia, congenital coagulopathies).

  2- Patients who received a blood product transfusion within the 7 days before MV initiation or during it.

  3- Patients with incomplete medical records or missing hematological data.

  4- Patients discharged or deceased within 24 hours of mechanical ventilation initiation.

  5- Patients who received Hematopoietic drugs during MV.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: the study will take place in Pediatric Intensive Care Unit (PICU) of (Assiut University Children's Hospital) with Pediatric patients aged 1 month to 18 years and Diagnosis of sepsis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
identify correlations between mechanical ventilation and hematological alterations in pediatric patients diagnosed with sepsis. | Baseline
  The primary outcome of the study is to identify correlations between mechanical ventilation and hematological alterations in pediatric patients diagnosed with sepsis. This includes assessing changes in blood parameters such as anemia, coagulation abnormalities, and inflammatory markers before and during mechanical ventilation.

SECONDARY OUTCOMES:
optimize patient management in critical care settings | Baseline
  optimize patient management in critical care settings by understanding the physiological effects of MV.
  * ICU and hospital mortality rates
  * Duration of mechanical ventilation in days
  * Length of ICU and hospital stay in days
  * Extubation success and reintubation rates
  * Incidence of ventilator-associated pneumonia (VAP)
  * Progression to acute respiratory distress syndrome (ARDS)
  * Need for renal replacement therapy during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Ismail lotfy mohamed, professor, Study Chair — Assiut University; mervat amin mahmoud, assistant professor, Study Director — Assiut University
Locations (1):
- Assiut University Children's Hospital, Asyut, Egypt

REFERENCES:
- [Background] Horak J, Martinkova V, Radej J, Matejovic M. Back to Basics: Recognition of Sepsis with New Definition. J Clin Med. 2019 Nov 1;8(11):1838. doi: 10.3390/jcm8111838. PMID 31683991
- [Background] Weiss SL, Peters MJ, Alhazzani W, Agus MSD, Flori HR, Inwald DP, Nadel S, Schlapbach LJ, Tasker RC, Argent AC, Brierley J, Carcillo J, Carrol ED, Carroll CL, Cheifetz IM, Choong K, Cies JJ, Cruz AT, De Luca D, Deep A, Faust SN, De Oliveira CF, Hall MW, Ishimine P, Javouhey E, Joosten KFM, Joshi P, Karam O, Kneyber MCJ, Lemson J, MacLaren G, Mehta NM, Moller MH, Newth CJL, Nguyen TC, Nishisaki A, Nunnally ME, Parker MM, Paul RM, Randolph AG, Ranjit S, Romer LH, Scott HF, Tume LN, Verger JT, Williams EA, Wolf J, Wong HR, Zimmerman JJ, Kissoon N, Tissieres P. Surviving Sepsis Campaign International Guidelines for the Management of Septic Shock and Sepsis-Associated Organ Dysfunction in Children. Pediatr Crit Care Med. 2020 Feb;21(2):e52-e106. doi: 10.1097/PCC.0000000000002198. PMID 32032273
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Fleischmann-Struzek C, Goldfarb DM, Schlattmann P, Schlapbach LJ, Reinhart K, Kissoon N. The global burden of paediatric and neonatal sepsis: a systematic review. Lancet Respir Med. 2018 Mar;6(3):223-230. doi: 10.1016/S2213-2600(18)30063-8. PMID 29508706